CLINICAL TRIAL: NCT06344091
Title: A Real World Study on Local Infiltration of Bupivacaine Liposome Injection for Acute Postoperative Pain After Pediatric Orthopedic Surgery
Brief Title: A Study of Bupivacaine Liposome Injection in Local Analgesia of Pediatric Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ZYWB-ZM-AHP-A-003
Record Dates: First submitted 2024-03-13; First posted 2024-04-03 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-06

CONDITIONS: Local Analgesia Via Infiltration

STUDY DESIGN:
Intervention Model Description: A single-arm study of liposomal bupivacaine injection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bupivacaine Liposome Injection (Experimental)
  Interventions: Drug: Bupivacaine Liposome Injection

INTERVENTIONS:
Drug: Bupivacaine Liposome Injection — Bupivacaine Liposome Injection 4 mg/kg (up to a maximum of 266 mg)

SUMMARY:
The study is being conducted to evaluate the safety and efficacy of bupivacaine liposome injection for local infiltration analgesia in pediatric orthopedic surgery in the real world.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects and guardians are willing to sign the informed consent.
2. Subjects undergoing orthopedic surgery under general anesthesia with expected cumulative incision length≥3cm.
3. 6 years old ≤ age ≤17 years old , Male or female.
4. ASA Physical Status Classification I-III.

Exclusion Criteria:

1. Subjects received liposomal bupivacaine or bupivacaine hydrochloride within the past 30 days;
2. Subjects with a history of immunodeficiency diseases (such as congenital immunodeficiency disease, AIDS or malignant tumors) or received immunosuppressants within 30 days;
3. Subjects with comorbid mental diseases (such as schizophrenia, depression, etc.) or difficult to communicate;
4. Subjects with a history of chronic pain or visceral pain;
5. Subjects with abnormal liver and kidney function;
6. Subjects with clinically significant abnormal heart rate or rhythm;
7. Subjects who are participating or planning to participate in any interventional clinical trial;
8. The investigators determined that other conditions were inappropriate for participation in this clinical trial.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 232 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2026-09-28 (Estimated); Study Completion 2026-10-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of Treatment Emergent Adverse events (TEAE) in the cardiac and nervous system | 0 minute to 14 days after administration
  Proportion of patients with any TEAE of cardiac or nervous system in MedDRA (Medical Dictionary for Regulatory Activities)

SECONDARY OUTCOMES:
The cumulative amount of opioids used in 0-24 hours, 24-48 hours, 48-72 hours and 0-72 hours after administration | 0 minute to 72 hours after administration
  Total consumption of opioids during 0-24 hours, 24-48 hours, 48-72 hours and 0-72 hours after administration.
Time to first rescue analgesia of opioid | 0 minute to 72 hours after administration
  Duration from administration to first use of opioid for rescue analgesia.
The proportion of patients who did not use rescue analgesia during 0-24 hours, 24-48 hours, 48-72 hours and 0-72 hours after administration | 0 minute to 72 hours after administration
  The proportion of patients who did not use rescue analgesia during 72 hours after administration.
The proportion of patients using patient-controlled intravenous analgesia (PCIA) | 0 minute to 72 hours after administration
  The proportion of patients who used patient-controlled intravenous analgesia (PCIA) during 0-72 hours after administration.
Pain intensity score at rest after administration for children aged 6 to 7 years | 0 minute to 72 hours after administration
  Wong Baker Faces Pain Scale Revision (FPS-R，0 indicates no pain and 10 indicates the most severe pain) was used for children aged 6 to 7 years at the time of 30minutes after awakening (including 30minutes), 6hours (±30minutes), 12hours (±30minutes), 18hours (±30minutes), 24hours (±30minutes), 36hours (±30minutes), 48hours (±30minutes) and 72hours (±30minutes).
Pain intensity score at rest after administration for children aged 8 years and older | 0 minute to 72 hours after administration
  Numercal Rating Scale (0 indicates no pain and 10 indicates the most severe pain) was used for children aged 8 years and older to assess the intensity of pain at the time of 30minutes after awakening (including 30minutes), 6hours (±30minutes), 12hours (±30minutes), 18hours (±30minutes), 24hours (±30minutes), 36hours (±30minutes), 48hours (±30minutes) and 72hours (±30minutes).
Pain intensity score on movement (or cough) after administration for children aged 6 to 7 years | 0 minute to 72 hours after administration
  Wong Baker Faces Pain Scale Revision (FPS-R，0 indicates no pain and 10 indicates the most severe pain) was used for children aged 6 to 7 years at the time of 30minutes after awakening (including 30minutes), 6hours (±30minutes), 12hours (±30minutes), 18hours (±30minutes), 24hours (±30minutes), 36hours (±30minutes), 48hours (±30minutes) and 72hours (±30minutes).
Pain intensity score on movement (or cough) after administration for children aged 8 years and older | 0 minute to 72 hours after administration
  Numercal Rating Scale (0 indicates no pain and 10 indicates the most severe pain) was used for children aged 8 years and older to assess the intensity of pain at the time of 30minutes after awakening (including 30minutes), 6hours (±30minutes), 12hours (±30minutes), 18hours (±30minutes), 24hours (±30minutes), 36hours (±30minutes), 48hours (±30minutes) and 72hours (±30minutes).
Length of Stay | up to 2 weeks
  The score of Post-Anesthetic Discharge Scoring System Scale (PADSS) was used to determine whether the patient could be discharged.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided